CLINICAL TRIAL: NCT07057466
Title: Prospective Evaluation of Artificial Intelligence-enhanced Electrocardiography for Detection of Structural Heart Disease
Brief Title: Prospective Evaluation of AI-ECG for SHD Detection
Acronym: AI-ECG-SHD
Status: Recruiting | Type: Observational
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Other Study IDs: 179372
Record Dates: First submitted 2025-06-26; First posted 2025-07-09 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Valvular Heart Disease Stenosis and Regurgitation (Diagnosis); Pulmonary Hypertension (Diagnosis); Heart Failure With Reduced Ejection Fraction (HFrEF; Diagnosis); Heart Failure With Preserved Ejection Fraction (HFpEF; Diagnosis)
Keywords: Artificial Intelligence; Machine Learning; Wearable Devices; Portable Devices; Heart Failure; Pulmonary Hypertension; Valvular Heart Disease; Echocardiography; Electrocardiography
MeSH Terms: conditions — Gastroesophageal Reflux; Disease; Hypertension, Pulmonary; Heart Failure; Heart Valve Diseases | interventions — Phlebotomy; pro-brain natriuretic peptide (1-76)

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood samples for NT-proBNP
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Echocardiography cohort: This cohort of patients will be attending for inpatient and outpatient transthoracic echocardiograms (TTEs) as part of their routine clinical care, having been referred by clinicians for various standard TTE indications, including investigation of symptoms such as breathlessness due to possible heart failure (HF), and screening for suspected valvular heart disease (VHD) and/or pulmonary hypertension (PH). These patients will have had no prior formal diagnosis of HF, VHD, and/or PH.
  Interventions: Other: Traditional 12-lead Electrocardiogram; Other: Apple Watch Series 4 Single-lead Electrocardiogram; Other: Eko Core 500 Digital Stethoscope 3-lead Electrocardiogram; Other: AliveCor KardiaMobile Single- and 6-lead Electrocardiogram
- N-terminal pro B-type natriuretic peptide subgroup: A subgroup of 203 patients, out of the total 590 patiets in the Echocardiography cohort, will be randomised to undergo blood tests and collection of serum N-terminal pro B-type natriuretic peptide (NT-proBNP).
  Interventions: Other: Traditional 12-lead Electrocardiogram; Other: Apple Watch Series 4 Single-lead Electrocardiogram; Other: Eko Core 500 Digital Stethoscope 3-lead Electrocardiogram; Other: AliveCor KardiaMobile Single- and 6-lead Electrocardiogram; Other: Phlebotomy for N-terminal pro-B-type natriuretic peptide

INTERVENTIONS:
Other: Traditional 12-lead Electrocardiogram — 12-lead ECG investigation is a standard, non-invasive diagnostic procedure used as an intervention to assess participants' cardiac electrical activity. For the purposes of this study, 12-lead ECGs will be collected for the application of AI-ECG models for the detection of HF, VHD, and/or PH and will not be used to inform or alter patients' standard NHS care.
Other: Apple Watch Series 4 Single-lead Electrocardiogram — Single-lead ECG taken using an Apple Watch Series 4 is a non-invasive, participant-initiated recording of cardiac electrical activity through a wearable device. While more limited than a 12-lead ECG, it can capture rhythm abnormalities-such as atrial fibrillation-and offers a convenient method for remote or continuous heart monitoring during the study. For the purposes of this study, single-lead ECGs will be collected for the application of AI-ECG models for the detection of HF, VHD, and/or PH and will not be used to inform or alter patients' standard NHS care.
Other: Eko Core 500 Digital Stethoscope 3-lead Electrocardiogram — Three-lead ECG recorded using the Eko CORE 500 digital stethoscope is a non-invasive, clinician-operated cardiac assessment tool that captures real-time electrical activity of the heart during auscultation. It provides enhanced diagnostic information compared to single-lead recordings, allowing detection of arrhythmias and signs of structural heart disease at the point of care, supporting integrated clinical and digital assessment. For the purposes of this study, 3-lead ECGs will be collected for the application of AI-ECG models for the detection of HF, VHD, and/or PH and will not be used to inform or alter patients' standard NHS care.
Other: AliveCor KardiaMobile Single- and 6-lead Electrocardiogram — A single- or 6-lead ECG recorded using the AliveCor KardiaMobile 6L device which is a portable, non-invasive method for capturing cardiac electrical activity. Operated by the participant or clinician, the device enables rapid rhythm assessment and detection of abnormalities such as atrial fibrillation. The 6-lead configuration offers more comprehensive data than single-lead recordings, supporting enhanced arrhythmia and conduction analysis in both in-clinic and remote settings. For the purposes of this study, single- and 6-lead ECGs will be collected for the application of AI-ECG models for the detection of HF, VHD, and/or PH and will not be used to inform or alter patients' standard NHS care.
Other: Phlebotomy for N-terminal pro-B-type natriuretic peptide — A minimally invasive biomarker assessment used to evaluate cardiac wall stress and function. Elevated levels can indicate the presence or severity of heart failure and other forms of structural heart disease, making it a valuable tool for diagnosis, risk stratification, and monitoring of cardiac status throughout the study period. For the purposes of this study, NT-proBNP will be collected to assess its accuracy at detecting HF, PH, and VHD with comparison with AI-ECG detections. The investigators will also evaluate the accuracy of AI-ECG detections combined with NT-pro-BNP, for detecting HF, VHD, and PH. The investigators will not be using NT-proBNP results to inform or alter patients' standard NHS care.
  Groups: N-terminal pro B-type natriuretic peptide subgroup

SUMMARY:
This study aims to improve the early detection of undiagnosed heart disease, which causes serious health issues, hospital admissions, and high healthcare costs. Researchers are exploring how artificial intelligence (AI) can analyse routine heart tests, called electrocardiograms (ECGs), to detect heart problems. These tests can be done using both traditional ECG machines and portable, wearable devices like smartwatches, making it easier for people to monitor their heart health at home.

While AI has shown promise using past data, this study will involve the collection of ECG data and subsequent testing of its accuracy in real-world settings to ensure it works well for both doctors and patients. The goal is to see if AI can identify conditions like heart muscle weakness, valve issues, and high lung pressure from the ECG data of patients. The researchers will also compare AI's detections with other blood tests commonly used to diagnose heart disease.

The AI models that will be used are being tested for research and validation purposes only. They will not be used for clinical decision-making or providing information to influence diagnosis, treatment, or patient care during the study. The AI outputs are not shared with clinicians and will have no impact on the care pathway.

This research will demonstrate if AI-powered ECG analysis - whether from traditional or portable devices - can provide a low-cost, non-invasive way to detect heart disease early and improve health assessments.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18-90 years
* No prior formal diagnosis of HF (including systolic and diastolic dysfunction), PH, or VHD
* Ability to provide informed consent

Exclusion Criteria:

* Severe arrhythmia or unstable cardiovascular disease
* Prior formal diagnosis of HF (including systolic and diastolic dysfunction), PH, or VHD
* Cardiac implantable electronic device in-situ, including a permanent pacemaker or implantable cardioverter defibrillator
* Involvement in current research or recent involvement in any research prior to recruitment

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This prospective observational cohort and validation study will recruit 590 unselected patients attending Chelsea and Westminster Hospital NHS Foundation Trust for routine echocardiography as part of their routine clinical care. Patients attending routine echocardiography who satisfy the inclusion and exclusion criteria will be approached before their echocardiography appointment to obtain informed consent to participate in the study.
Sampling Method: Non-Probability Sample
Enrollment: 590 (Estimated)
Dates: Start 2025-11-04 (Actual); Primary Completion 2027-05-03 (Estimated); Study Completion 2027-08-02 (Estimated)

PRIMARY OUTCOMES:
AI-ECG model classification performance for detection of structural heart disease (SHD) | From enrolment to end of patient's study visit (up to 1 hour)
  AI-ECG model classification performance for HF, PH, and VHD, will be assessed for all ECG modalities (single-, 3-, 6-, and 12-lead ECGs) using the area under the receiver operating characteristic (AUROC; pre-defined threshold).

SECONDARY OUTCOMES:
Additional AI-ECG performance metrics for detection of SHD | From enrolment to end of patient's study visit (up to 1 hour)
  Secondary performances measures will include sensitivity, specificity, negative predictive value (NPV), positive predictive value (PPV) and F1 score for all ECG modalities.
NT-proBNP performance metrics for detection of SHD | From enrolment to end of patient's study visit (up to 1 hour)
  performances measures will include area under the receiver operating characteristic (AUROC; pre-defined threshold), sensitivity, specificity, negative predictive value (NPV), positive predictive value (PPV) and F1 score for all ECG modalities.
Combined AI-ECG and NT-proBNP performance analysis for detection of SHD | From enrolment to end of patient's study visit (up to 1 hour)
  NT-proBNP and AI-ECG predictions will be combined in a logistic regression model to assess the performance of a combined approach.

CONTACTS AND LOCATIONS:
Locations (2):
- United Kingdom (2):
  - Chelsea and Westminster Hospital, London
  - West Middlesex University Hospital, London

IPD SHARING:
Plan to Share IPD: No